CLINICAL TRIAL: NCT04824963
Title: Analysis of Related Factors Affecting the Secondary Implantation of IOLs in Congenital Cataract
Brief Title: Analysis of Related Factors Affecting the Secondary Implantation of Intraocular Lens in Congenital Cataract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: WDD-secondary implantation
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-03

CONDITIONS: Congenital Cataract
Keywords: secondary implantation; ciliary sulcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ocular biometric parameters of the children with congenital cataract including preoperative pupil diameter, corneal diameter, axial length, anterior and posterior capsule size, iris adhesion. And then analysis whether the preoperative parameters were correlated with the implantation site of secondary implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as congenital cataract without lens after surgery
* Secondare IOLs implantation surgery was performed in Eye hospital of Wenzhou Medical University

Exclusion Criteria:

* Suffers from uveitis, glaucoma and other ocular diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Congenital cataract patient accepted secondary IOLs implantation at Eye hospital of Wenzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
pupil diameter | Before lens implantation
  preoperative pupil diameter size
posterior capsule diameter | Before lens implantation
  preoperative posterior capsule diameter size

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China